CLINICAL TRIAL: NCT05136755
Title: NMDA Modulation in Antidepressant Nonresponders With Major Depressive Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH110-REC3-123
Record Dates: First submitted 2021-11-16; First posted 2021-11-29 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Antidepressant nonresponders; NMDA
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMDAE (Experimental): An NMDA enhancer
  Interventions: Drug: NMDAE
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Cap

INTERVENTIONS:
Drug: NMDAE — Use of an NMDA enhancer for the treatment of antidepressant nonresponders with MDD
  Arms: NMDAE
Drug: Placebo Cap — Use of placebo as a comparator
  Arms: Placebo

SUMMARY:
Most of the current antidepressants for major depressive disorder (MDD) are based upon the monoamine hypothesis which cannot fully explain the etiology of depression. NMDA hypofunction has been implicated in the pathophysiology of depression. This study aims to examine the efficacy and safety of an NMDA enhancer (NMDAE) in the treatment of antidepressant nonresponders with MDD.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a multi-factorial disorder. Most of the current antidepressants are based upon the monoamine hypothesis which cannot fully explain the etiology of depression. Many patients respond poorly to antidepressants and suffer from side effects. NMDA hypofunction has been implicated in the pathophysiology of depression. MDD is often associated with cognitive deficits which are not necessarily recovered by current antidepressants. The NMDA receptor regulates synaptic plasticity, memory, and cognition. Therefore, this study aims to examine the efficacy and safety as well as cognitive function improvement of NMDAE in the treatment of antidepressant nonresponders with MDD. The investigators will enroll a total of 50 antidepressant nonresponders with MDD. All patients, continuing their originally ongoing treatment throughout the study period, will be randomly assigned into either of two treatment groups: NMDAE or placebo. We will biweekly measure clinical performances using 17-item Hamilton Rating Scale for Depression, Global Assessment of Function, Perceived Stress Scale, Visual Analogue Scale for pain, Clinical Global Impression, and side effects. Quality of life and cognitive functions will be assessed at baseline and at endpoint of treatment.

The efficacies of NMDAE and placebo will be compared. Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSM-5 (American Psychiatric Association) diagnosis of MDD
* Have failed to respond to at least one antidepressant with adequate dosage and treatment duration
* Their original treatments should have been unchanged for at least 8 weeks. Some treatment-resistant patients (that is, having failed to respond to at least two different classes of antidepressants) who have started to refuse any antidepressant by themselves due to previous failure experience are also allowed, if they have already been antidepressant-free for at least 2 weeks
* 17-item Hamilton Rating Scale for Depression total score ≥ 18
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* Current substance abuse or history of substance dependence in the past 6 months
* History of epilepsy, head trauma, stroke or other serious medical or neurological illness which may interfere with the study
* Bipolar disorder, schizophrenia or other psychotic disorder
* Moderate-severe suicidal risks
* Severe cognitive impairment
* Initiating or stopping formal psychotherapy within six weeks prior to enrollment
* A history of previously received electroconvulsive therapy
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Rating Scale for Depression | week 0, 2, 4, 6, 8
  Assessment of depressive symptoms Minimum value: 0, maximum value:52, the higher scores mean a worse outcome.
Change in Global Assessment of Functioning | Week 0, 2, 4, 6, 8
  Assessment of global improvement. Minimum value: 1, maximum value:100, the higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change Change in Perceived Stress Scalein Perceived Stress Scale | week 0, 2, 4, 6, 8
  Assessment of stress and anxiety symptoms Minimum value: 0, maximum value:56, the higher scores mean a worse outcome.
Visual Analogue Scale for pain | week 0, 2, 4, 6, 8
  Assessment of pain Minimum value: 0, maximum value:10, the higher scores mean a worse outcome.
Clinical Global Impression | week 0, 2, 4, 6, 8
Quality of life (SF-36) | week 0, 8
Visual Continuous Performance Test | week 0, 8
  Assessment of sustained attention
Wisconsin Card Sorting Test | week 0, 8
  Assessment of abstract and shift set
Logical Memory Test of the Wechsler Memory Scale | week 0, 8
  Assessment of episodic memory
Digit Span | week 0, 8
  Assessment of verbal working memory
Spatial Span | week 0, 8
  Assessment of nonverbal working memory
Category Fluency | week 0, 8
  Assessment of speed of processing
Trail Marking A | week 0, 8
  Assessment of speed of processing
WAIS-III Digit Symbol-Coding | week 0, 8
  Assessment of speed of processing
Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) V2.0 | week 0, 8
  Assessment of social cognition

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan